CLINICAL TRIAL: NCT01751542
Title: Mindfulness and Acceptance Group Therapy for Substance Use
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8888-B
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Substance Use Disorder
MeSH Terms: conditions — Substance-Related Disorders | interventions — Mindfulness; Residential Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness + residential treatment (Experimental): Mindfulness and Acceptance Group Therapy + residential treatment
  Interventions: Behavioral: Mindfulness + Residential Treatment
- Residential Treatment (Active Comparator): Residential treatment alone
  Interventions: Behavioral: Residential treatment alone

INTERVENTIONS:
Behavioral: Mindfulness + Residential Treatment
  Arms: Mindfulness + residential treatment
Behavioral: Residential treatment alone
  Arms: Residential Treatment

SUMMARY:
Randomized clinical trial comparing standard residential substance abuse treatment to standard residential treatment plus Mindfulness and Acceptance Group Therapy for substance use.

ELIGIBILITY:
Inclusion Criteria:

* participating in inpatient substance use treatment at treatment facility

Exclusion Criteria:

* psychosis and mental impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Substance use after discharge from treatment | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tenneessee & Cornerstone of Recovery, Knoxville, Tennessee, United States